CLINICAL TRIAL: NCT01380886
Title: Growth and Tolerance of Young Infants Fed Infant Formulas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK92
Record Dates: First submitted 2011-06-16; First posted 2011-06-27 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Infant Newborn

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infant formula, alternate protein source (Experimental): Experimental infant formula with alternate protein source
  Interventions: Other: experimental infant formula with alternate protein source
- Infant formula powder (Active Comparator): Infant formula powder
  Interventions: Other: Infant formula powder

INTERVENTIONS:
Other: experimental infant formula with alternate protein source — experimental infant formula to be fed ad libitum
  Arms: Infant formula, alternate protein source
Other: Infant formula powder — powdered infant formula to be fed ad libitum
  Arms: Infant formula powder

SUMMARY:
This is a randomized, multi-center, double blind, parallel study to compare growth and tolerance of healthy term infants fed either control or experimental infant formula.

ELIGIBILITY:
Inclusion Criteria:

* healthy infant
* full term
* birth weight > 2490 g
* 0 to 8 days of age
* parent/physician agree to not use medications affecting tolerance/growth
* parent agrees to sole source feeding of study formula
* parent agrees to not use vitamin/mineral supplements
* parent has signed consent/HIPAA authorization

Exclusion Criteria:

* any maternal, fetal, or infant history affecting growth and tolerance
* participation in any other study not preapproved by Abbott

Max Age: 8 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 209 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Weight gain | 119 days

SECONDARY OUTCOMES:
gastrointestinal tolerance | 119 days
  Stool characteristics, number of stools per day, and number of feedings associated with spit up or vomit
Anthropometric variables | 119 days
  Length gain per day and head circumference gain per day

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Borschel, PhD, Study Chair — Abbott Nutrition
Locations (12):
- United States (12):
  - Norwich Pediatric Group, PC, Norwich, Connecticut
  - SCORE Physician Alliance, LLC, St. Petersburg, Florida
  - Northpoint Pedicatrics, LLC, Indianapolis, Indiana
  - Springs Medical Research, LLC, Owensboro, Kentucky
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Cary Pediatric Center, Cary, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio Pediatric Research Association, INC., Huber Heights, Ohio
  - Institute of Clinical Research, Mayfield Heights, Ohio
  - The Cleveland Pediatric Research Center, Parma, Ohio
  - Sanford Clinic Family Medicine, Sioux Falls, South Dakota
  - DCOL Center for Clinical Research, Longview, Texas